CLINICAL TRIAL: NCT04321694
Title: Expanded Access for KHK2455
Status: No longer available | Type: Expanded Access
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: University of New Mexico Cancer Center (Other)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: Expanded Access for KHK2455
Record Dates: First submitted 2020-01-21; First posted 2020-03-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — mogamulizumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: KHK2455
  Other Names: Mogamulizumab

SUMMARY:
This is an expanded access program for eligible participants. This program is designed to provide access to KHK2455 in combination with Mogamulizumab prior to the approval by the local regulatory agency. A medical doctor must decide whether the potential benefit outweighs the risk of receiving this investigational therapy based on the individual patients medical history and eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult